CLINICAL TRIAL: NCT03973489
Title: Effects of Genotype on Resting State Connectivity During Methamphetamine Administration
Acronym: MATAAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Hoffman, PhD, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17932
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Methamphetamine-dependence
Keywords: Methamphetamine
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects will be grouped into either the CV or WT group. Neither they nor the researchers will know which group they are in. In addition, subjects will be randomly assigned to receive drug then placebo or placebo than drug. Neither researchers or subjects will know in which order they will receive drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Wild Type (WT) MUD Group (Experimental): Wild Type (WT) Group: individuals who are WT for the TAAR1 gene
  Interventions: Behavioral: Magnetic resonance imaging (MRI); Drug: Methamphetamine Hydrochloride Tablets; Drug: Placebo oral tablet
- Common Variant (CV) MUD Group (Experimental): Common Variant (CV) Group: individuals who are hetero-or homozygous for the valine codon occurring at amino acid position 288, designated V288V, SNP on the TAAR1 gene
  Interventions: Behavioral: Magnetic resonance imaging (MRI); Drug: Methamphetamine Hydrochloride Tablets; Drug: Placebo oral tablet
- Wild Type (WT) Healthy Control Group (Experimental): Wild Type (WT) Group: individuals who are WT for the TAAR1 gene
  Interventions: Behavioral: Magnetic resonance imaging (MRI); Drug: Methamphetamine Hydrochloride Tablets; Drug: Placebo oral tablet
- Common Variant (CV) Healthy Control Group (Experimental): Common Variant (CV) Group: individuals who are hetero-or homozygous for the V288V SNP on the TAAR1 gene
  Interventions: Behavioral: Magnetic resonance imaging (MRI); Drug: Methamphetamine Hydrochloride Tablets; Drug: Placebo oral tablet

INTERVENTIONS:
Behavioral: Magnetic resonance imaging (MRI) — On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
Drug: Methamphetamine Hydrochloride Tablets — Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Other Names: Desoxyn
Drug: Placebo oral tablet — Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.

SUMMARY:
Addiction to methamphetamine (MA) is a serious health problem in the United States. Right now, there are no medically approved treatments for MA dependence. More research is needed to understand how MA affects the brain and to eventually develop medical interventions for MA addiction. The purpose of the study is to learn more about how MA use affects the brain by investigating a receptor in the brain called trace amine-associated receptor 1 (TAAR1). The investigators are hoping to find out if individuals with certain versions of the brain receptor react differently when given MA. The TAAR1 receptor has two prevalent genetic variations due to a single nucleotide polymorphism. These are the wild type (WT) and a common variant (CV). Preliminary studies have shown that these variants produce different connectivity (resting state functional connectivity or RSFC) in the brains of individuals with MA use disorder (MUD), specifically that individuals with the CV genotype exhibit lower RSFC than WT. In this study, MA will be administered to individuals with MA use disorder and healthy controls in order to:

1. Determine the influence of CV vs. WT genotype on RSFC and craving in individuals with chronic MUD and healthy controls.
2. Determine the effect of acute methamphetamine or placebo administration on the interaction of CV vs WT genotype on RSFC, craving, cognitive control, attention and subjective experience in MUD and healthy controls.

DETAILED DESCRIPTION:
This proposal will determine the effect of a common variant (CV) synonymous single nucleotide polymorphism (SNP) of the gene for the human trace amine associated receptor 1 (TAAR1) on the neural and behavioral response of subjects with methamphetamine (MA) use disorder (MUD) and healthy control subjects to acute MA administration. The SNP (rs8192620 on human Genome Reference Consortium Human Build 38 patch release 7 chromosome 6 at 132,645,140 bp in htaar1, allelic frequency 22%) results from a change of adenine to guanine in a valine codon occurring at amino acid position 288 (V288V). MA is a potent agonist at the TAAR1 receptor, in addition to its actions at the dopamine transporter and the vesicular monoamine transporter. In rodents, a decrease in TAAR1 expression or non-functional TAAR1 receptor is associated with an increase in striatal dopamine (DA) signaling.

The scientific premise of this project is based on 1) preliminary findings that support a model that the CV alters RSFC of the striatum, a dopaminergic terminal region, and associated behavior in chronic MUD, 2) published reports that delineate the effect of TAAR1 on DA signaling and 3) preclinical evidence that TAAR1 influences sensitivity to rewarding and aversive effects of MA.

Furthermore, this proposal will address questions that have important implications for understanding and treating patients with MUD, as the TAAR1 receptor is implicated in MA self-administration. As an allele of the murine TAAR1 gene associated with an inactive receptor leads to increased MA intake in homozygotes, it is critically important to study the feasibility of exploiting human variant htaar1.

The investigators propose a model based on this premise that makes testable predictions about the interaction of the CV with chronic and acute MA administration in MUD. The investigators' preliminary data show that the CV causes over-expression of TAAR1 in cell culture. Stimulation of the TAAR1 receptor decreases dopaminergic signaling in mesocorticolimbic and corticostriatal networks. The investigators propose that this effect in conjunction with chronic MA use causes neuroadaptations that result in the increased striato- and corticolimbic RSFC as well as increased drug craving observed in MUD subjects with the CV. The investigators can indirectly test the hypothesis of decreased DA release due to ever-expression via MA administration. The effect of acute MA administration on RSFC in humans is not known but acute administration of S-amphetamine and methylphenidate reduce RSFC in salience attribution and default mode networks presumably via increased DA release. Stimulation of over-expressed TAAR1 should blunt this effect in CV carrying individuals compared to WT. There are no published reports on neural effects of the interaction between either chronic or acute MA administration and htaar1 genotype in humans, therefore this proposal represents a unique opportunity to determine whether the RSFC response to acute MA administration in humans is mediated by genotype.

ELIGIBILITY:
Criteria for Inclusion:

[All groups]

* 18 to 55 years old
* Homozygous or heterozygous for the human TAAR1 (hTAAR1) V288V genotype or wild type for hTAAR1 (determined during screening visit "Visit 1")

[Meth use group]

* Subjects must have a positive urine drug screen for methamphetamine during visit one
* Meets current criteria for methamphetamine use disorder
* Subjects should have been using at least 100mg of methamphetamine (not prescribed), 5 days per week for at least one year
* Abstinent from methamphetamine for 24 hours on days of scans

[Healthy volunteer group]

- At least one exposure to a stimulant, either recreational or prescribed

Criteria for Exclusion:

[All groups]

* Allergies to stimulants or hypersensitivity to taking a stimulant in the past
* Diagnosis of a psychotic or mood disorder
* Self-reported claustrophobia
* Women who are pregnant or breast-feeding
* Intoxicated on study days
* Clinically significant neurological, cardiovascular, endocrine, renal, hepatic or systemic disease that could compromise safe participation or confound outcomes (including hepatitis C, HIV, severe anemia, or liver disease)
* History of glaucoma
* Metal in the body which is contraindicated for MRI or would compromise image quality
* Current prescription use of stimulants, anti-psychotic drugs or anti-Parkinson's drugs
* Use of monoamine oxidase inhibitors within 14 days
* Use of serotonin reuptake inhibiters, serotonin norepinephrine reuptake inhibiters, triptans, tricyclic antidepressants, Fentanyl, lithium, tramadol, tryptophan, buspirone , St. John's Wort, insulin, phenothiazines, guanethidine, acidifying/alkalinizing agents, CYP2D6 inhibitors, proton pump inhibitors

[Meth use group]

* Positive urine drug screen at any point during the study (except for meth or marijuana)
* History of any severe substance use disorders within the last 5 years, except for methamphetamine use disorder or tobacco use disorder

[Healthy volunteer group]

* History of any severe substance use disorders within the last 5 years except tobacco use disorder
* Positive urine drug screen at any point in the study (except for marijuana or for verified medical reasons)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hoffman, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wild Type (WT) MUD Group: Methamphetamine First, Then Placebo; Wild Type (WT) MUD Group: Placebo First, Then Methamphetamine; Wild Type (WT) Healthy Control Group: Methamphetamine First, Then Placebo; Wild Type (WT) Healthy Control Group: Placebo First, Then Methamphetamine: Wild Type (WT) Group: individuals who are WT for the TAAR1 gene
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- Common Variant (CV) MUD Group: Methamphetamine First, Then Placebo; Common Variant (CV) MUD Group: Placebo First, Then Methamphetamine: Common Variant (CV) Group: individuals who are hetero-or homozygous for the valine codon occurring at amino acid position 288 (V288V) single nucleotide polymorphism (SNP) on the TAAR1 gene
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- Common Variant (CV) Healthy Control Group: Methamphetamine First, Then Placebo; Common Variant (CV) Healthy Control Group: Placebo First, Then Methamphetamine: Common Variant (CV) Group: individuals who are hetero-or homozygous for the V288V SNP on the TAAR1 gene
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
Period: First Intervention (1 Day)
Arm/Group | Wild Type (WT) MUD Group: Methamphetamine First, Then Placebo | Wild Type (WT) MUD Group: Placebo First, Then Methamphetamine | Common Variant (CV) MUD Group: Methamphetamine First, Then Placebo | Common Variant (CV) MUD Group: Placebo First, Then Methamphetamine | Wild Type (WT) Healthy Control Group: Methamphetamine First, Then Placebo | Wild Type (WT) Healthy Control Group: Placebo First, Then Methamphetamine | Common Variant (CV) Healthy Control Group: Methamphetamine First, Then Placebo | Common Variant (CV) Healthy Control Group: Placebo First, Then Methamphetamine
Started | 4 | 3 | 2 | 5 | 4 | 4 | 2 | 2
Completed | 4 | 3 | 2 | 5 | 4 | 4 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 3 Days)
Arm/Group | Wild Type (WT) MUD Group: Methamphetamine First, Then Placebo | Wild Type (WT) MUD Group: Placebo First, Then Methamphetamine | Common Variant (CV) MUD Group: Methamphetamine First, Then Placebo | Common Variant (CV) MUD Group: Placebo First, Then Methamphetamine | Wild Type (WT) Healthy Control Group: Methamphetamine First, Then Placebo | Wild Type (WT) Healthy Control Group: Placebo First, Then Methamphetamine | Common Variant (CV) Healthy Control Group: Methamphetamine First, Then Placebo | Common Variant (CV) Healthy Control Group: Placebo First, Then Methamphetamine
Started | 4 | 3 | 2 | 5 | 4 | 4 | 2 | 2
Completed | 2 | 3 | 2 | 3 | 1 | 4 | 1 | 2
Not Completed | 2 | 0 | 0 | 2 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Too much motion in scanner | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Wild Type (WT) MUD Group: Methamphetamine First, Then Placebo | Wild Type (WT) MUD Group: Placebo First, Then Methamphetamine | Common Variant (CV) MUD Group: Methamphetamine First, Then Placebo | Common Variant (CV) MUD Group: Placebo First, Then Methamphetamine | Wild Type (WT) Healthy Control Group: Methamphetamine First, Then Placebo | Wild Type (WT) Healthy Control Group: Placebo First, Then Methamphetamine | Common Variant (CV) Healthy Control Group: Methamphetamine First, Then Placebo | Common Variant (CV) Healthy Control Group: Placebo First, Then Methamphetamine
Started | 2 | 3 | 2 | 3 | 1 | 4 | 1 | 2
Completed | 2 | 3 | 2 | 2 | 1 | 4 | 1 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Common Variant (CV) MUD Group; Common Variant (CV) Healthy Control Group: Common Variant (CV) Group: individuals who are hetero-or homozygous for the V288V SNP on the TAAR1 gene
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- Total: Total of all reporting groups
Arm/Group | Wild Type (WT) MUD Group | Common Variant (CV) MUD Group | Wild Type (WT) Healthy Control Group | Common Variant (CV) Healthy Control Group | Total
Number analyzed (Participants) | 7 | 7 | 8 | 4 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 8 | 4 | 26
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 2 | 11
  Male | 6 | 3 | 4 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 5 | 8 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 7 | 4 | 6 | 4 | 21
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity During Resting State Magnetic Resonance Imaging (MRI)
Description: Pearson correlation coefficient (r) was used to calculate cortico-striatal and intra-striatal functional connectivity during resting state. These r values were then converted into Fisher's Z-scores using the transformation: z = arctanh(r) = 0.5*ln((1+r)/(1-r)). Fisher's Z-transformation linearizes Pearson correlations and allows for statistical analysis. The Z-scores represent the strength and direction of functional connectivity between brain regions. A Z-score of 0 represents the population mean for functional connectivity between brain regions. Larger Z-scores indicate stronger connectivity (potentially indicating greater activation or association), while smaller (negative) Z-scores indicate weaker connectivity, which could suggest reduced synchronization or disrupted brain function. Z-scores above or below ±1 standard deviation from the mean may indicate notable deviations from the expected connectivity patterns in the population.
Time Frame: 1 hour prior to and 1.5 hours post study drug administration on visits 2 and visit 3 (randomized to placebo or methamphetamine; washout period between visit 2 and 3 was at least 3 days)
Population: Participants were excluded from further analyses if they did not complete pre and post imaging outcome measures during visit. Placebo and methamphetamine administration include individuals who completed the respective visit at either the first or second intervention.
Measure: Mean (Standard Deviation); unit: Fisher's Z-score
Groups:
- MUD Group, CV Genotype, Pre Placebo Administration: Individuals with Methamphetamine Use Disorder (MUD) and Common Variant (CV) of the TAAR1 genotype prior to receiving placebo during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, CV Genotype, Post Placebo Administration: Individuals with Methamphetamine Use Disorder (MUD) and Common Variant (CV) of the TAAR1 genotype after placebo administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, WT Genotype, Pre Placebo Administration: Individuals with Methamphetamine Use Disorder (MUD) and Wild Type (WT) variant of the TAAR1 genotype prior to receiving placebo during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, WT Genotype, Post Placebo Administration: Individuals with Methamphetamine Use Disorder (MUD) and Wild Type (WT) variant of the TAAR1 genotype after placebo administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, CV Genotype, Pre Methamphetamine Administration: Individuals with Methamphetamine Use Disorder (MUD) and Common Variant (CV) of the TAAR1 genotype prior to receiving methamphetamine during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, CV Genotype, Post Methamphetamine Administration: Individuals with Methamphetamine Use Disorder (MUD) and Common Variant (CV) of the TAAR1 genotype after methamphetamine administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, WT Genotype, Pre Methamphetamine Administration: Individuals with Methamphetamine Use Disorder (MUD) and Wild Type (WT) variant of the TAAR1 genotype prior to receiving methamphetamine during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- MUD Group, WT Genotype, Post Methamphetamine Administration: Individuals with Methamphetamine Use Disorder (MUD) and Wild Type (WT) variant of the TAAR1 genotype after methamphetamine administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, CV Genotype, Pre Placebo Administration: Healthy Controls (HC) with no substance use disorders and Common Variant (CV) of the TAAR1 genotype prior to receiving placebo during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, CV Genotype, Post Placebo Administration: Healthy Controls (HC) with no substance use disorders and Common Variant (CV) of the TAAR1 genotype after placebo administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, WT Genotype, Pre Placebo Administration: Healthy Controls (HC) with no substance use disorders and Wild Type (WT) variant of the TAAR1 genotype prior to receiving placebo during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, WT Genotype, Post Placebo Administration: Healthy Controls (HC) with no substance use disorders and Wild Type (WT) variant of the TAAR1 genotype after placebo administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, CV Genotype, Pre Methamphetamine Administration: Healthy Controls (HC) with no substance use disorders and Common Variant (CV) of the TAAR1 genotype prior to receiving methamphetamine during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, CV Genotype, Post Methamphetamine Administration: Healthy Controls (HC) with no substance use disorders and Common Variant (CV) of the TAAR1 genotype after methamphetamine administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, WT Genotype, Pre Methamphetamine Administration: Healthy Controls (HC) with no substance use disorders and Wild Type (WT) variant of the TAAR1 genotype prior to receiving methamphetamine during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
- HC Group, WT Genotype, Post Methamphetamine Administration: Healthy Controls (HC) with no substance use disorders and Wild Type (WT) variant of the TAAR1 genotype after methamphetamine administration during visit.
  Magnetic resonance imaging (MRI): On visits 2 and 3, subjects will undergo a baseline MRI scan approximately 1 hour after the start of each visit followed by drug administration (placebo or MA) and a second scan 1.5 hours after that.
  Methamphetamine Hydrochloride Tablets: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits. Participants will receive the following doses of methamphetamine hydrochloride in accordance with their weight: if weight is between 50-60 kg, 15 mg dose of methamphetamine hydrochloride will be administered. Similarly, for 60-80 kg, 20 mg dose; 80-100 kg, 25 mg dose; and 100+ kg, 30 mg dose.
  Placebo oral tablet: Study participants will receive an oral dose of methamphetamine hydrochloride on one of two scan days and an identical looking placebo in tablet form on the other scan day. Drug type will be randomized between the two visits.
Arm/Group | MUD Group, CV Genotype, Pre Placebo Administration | MUD Group, CV Genotype, Post Placebo Administration | MUD Group, WT Genotype, Pre Placebo Administration | MUD Group, WT Genotype, Post Placebo Administration | MUD Group, CV Genotype, Pre Methamphetamine Administration | MUD Group, CV Genotype, Post Methamphetamine Administration | MUD Group, WT Genotype, Pre Methamphetamine Administration | MUD Group, WT Genotype, Post Methamphetamine Administration | HC Group, CV Genotype, Pre Placebo Administration | HC Group, CV Genotype, Post Placebo Administration | HC Group, WT Genotype, Pre Placebo Administration | HC Group, WT Genotype, Post Placebo Administration | HC Group, CV Genotype, Pre Methamphetamine Administration | HC Group, CV Genotype, Post Methamphetamine Administration | HC Group, WT Genotype, Pre Methamphetamine Administration | HC Group, WT Genotype, Post Methamphetamine Administration
Number analyzed (Participants) | 7 | 7 | 5 | 5 | 4 | 4 | 7 | 7 | 3 | 3 | 5 | 5 | 4 | 4 | 8 | 8
Fisher's Z-score
  Cortico striatal | 0.91 (0.96) | 0.52 (0.29) | 0.54 (0.5) | 0.32 (0.14) | 0.34 (0.22) | 0.49 (0.29) | 0.21 (0.33) | 0.58 (0.36) | 0.09 (0.04) | 0.14 (0.15) | 0.18 (0.09) | 0.15 (0.1) | 0.142 (0.09) | 0.101 (0.56) | 0.010 (0.10) | 0.164 (0.09)
  Intra-striatal | 0.36 (0.06) | 0.3 (0.09) | 0.25 (0.15) | 0.20 (0.14) | 0.19 (0.11) | 0.25 (0.10) | 0.23 (0.84) | 0.10 (0.08) | 0.25 (0.81) | 0.24 (0.18) | 0.35 (0.14) | 0.31 (0.09) | 0.192 (0.09) | 0.19 (0.32) | 0.26 (0.16) | 0.17 (0.21)

2. Primary Outcome: Euphoria Effects of Study Drug
Description: The Morphine Benzedrine group (MBG) scale is a subscale of the Addiction Research Center Inventory (ARCI-49), a 49 item questionnaire consisting of true/false items, which measures the euphoric effects of the study drug. The MBG scale ranges from 0-16 with higher numbers indicating more euphoria. The questionnaire was administered every hour for four hours following study drug administration and the highest score during this time is considered the post drug administration score.
Time Frame: 2.5 hours prior to and between 1-4 hours post study drug administration on visits 2 and visit 3 (randomized to placebo or methamphetamine; washout period between visit 2 and 3 was at least 3 days)
Population: Participants were excluded from further analyses if they did not complete all pre and post imaging measures during visit. Placebo and methamphetamine administration include individuals who completed the respective visit at either the first or second intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MUD Group, CV Genotype, Pre Placebo Administration | MUD Group, CV Genotype, Post Placebo Administration | MUD Group, WT Genotype, Pre Placebo Administration | MUD Group, WT Genotype, Post Placebo Administration | MUD Group, CV Genotype, Pre Methamphetamine Administration | MUD Group, CV Genotype, Post Methamphetamine Administration | MUD Group, WT Genotype, Pre Methamphetamine Administration | MUD Group, WT Genotype, Post Methamphetamine Administration | HC Group, CV Genotype, Pre Placebo Administration | HC Group, CV Genotype, Post Placebo Administration | HC Group, WT Genotype, Pre Placebo Administration | HC Group, WT Genotype, Post Placebo Administration | HC Group, CV Genotype, Pre Methamphetamine Administration | HC Group, CV Genotype, Post Methamphetamine Administration | HC Group, WT Genotype, Pre Methamphetamine Administration | HC Group, WT Genotype, Post Methamphetamine Administration
Number analyzed (Participants) | 7 | 7 | 5 | 5 | 4 | 4 | 7 | 7 | 3 | 3 | 5 | 5 | 4 | 4 | 8 | 8
score on a scale | 2.9 (2.0) | 6.0 (3.6) | 3.0 (2.2) | 5.2 (3.7) | 1.3 (1.5) | 4.8 (1.5) | 3.3 (2.5) | 6.0 (3.5) | 1.7 (0.6) | 3.0 (2.0) | 4.6 (3.4) | 5.8 (4.0) | 2.3 (2.5) | 8.8 (4.9) | 3.0 (1.7) | 10.9 (4.1)

3. Primary Outcome: Craving Assessed With the Stimulant Craving Questionnaire (STCQ)
Description: Current craving for methamphetamine was assessed using the Stimulant Craving Questionnaire (STCQ), which is a 10-item self-report measure that uses a seven-point scale, with answers ranging from 0 ("strongly disagree") to 6 ("strongly agree"). A composite score was computed by averaging the responses for all 10 items after reverse scoring items 4 and 7. Scores range from 0 to 6 with higher scores representing higher craving for methamphetamine.
Time Frame: 2 hours prior to and 3 hours post study drug administration on visits 2 and visit 3 (randomized to placebo or methamphetamine; washout period between visit 2 and 3 was at least 3 days)
Population: Participants were excluded from further analyses if they did not complete pre and post imaging measures during visit. Placebo and methamphetamine administration include individuals who completed the respective visit at either the first or second intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MUD Group, CV Genotype, Pre Placebo Administration | MUD Group, CV Genotype, Post Placebo Administration | MUD Group, WT Genotype, Pre Placebo Administration | MUD Group, WT Genotype, Post Placebo Administration | MUD Group, CV Genotype, Pre Methamphetamine Administration | MUD Group, CV Genotype, Post Methamphetamine Administration | MUD Group, WT Genotype, Pre Methamphetamine Administration | MUD Group, WT Genotype, Post Methamphetamine Administration | HC Group, CV Genotype, Pre Placebo Administration | HC Group, CV Genotype, Post Placebo Administration | HC Group, WT Genotype, Pre Placebo Administration | HC Group, WT Genotype, Post Placebo Administration | HC Group, CV Genotype, Pre Methamphetamine Administration | HC Group, CV Genotype, Post Methamphetamine Administration | HC Group, WT Genotype, Pre Methamphetamine Administration | HC Group, WT Genotype, Post Methamphetamine Administration
Number analyzed (Participants) | 7 | 7 | 5 | 5 | 4 | 4 | 7 | 7 | 3 | 3 | 5 | 5 | 4 | 4 | 8 | 8
units on a scale | 3.9 (1.4) | 3.2 (1.4) | 2.7 (1.3) | 2.3 (1.2) | 4.3 (1.2) | 4.3 (1.3) | 1.7 (1.5) | 2.1 (1.2) | 0 (0) | 0.2 (0.3) | 0.3 (0.4) | 0.2 (0.4) | 0.2 (0.3) | 0.4 (0.6) | 0.1 (0.2) | 0.2 (0.3)

4. Primary Outcome: Cognitive Function
Description: Two computer tests were administered to measure how each medication intervention effects cognitive functioning. The tests administered included the Rapid Visual Information Processing Task (RVIPT), a 6 minute test of sustained attention in which participants are requested to detect target sequences of digits and the Digit Symbol Substitution Task (DSST), a 2 minute test of psychomotor speed and sustained attention consisting of digit-symbol pairs followed by a list of digits where the subject identifies the symbol that corresponds to each digit as fast as possible. The number of correct responses within the allowed time is measured. Higher scores on both tasks indicate better performance.
Time Frame: as for outcome 3
Population: Participants were excluded from further analyses if they did not complete pre and post imaging measures during visit. Placebo and methamphetamine administration include individuals who completed the respective visit at either the first or second intervention. One participant (MUD, CV, post placebo administration) did not complete the final set of data but did complete both imaging measures.
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | MUD Group, CV Genotype, Pre Placebo Administration | MUD Group, CV Genotype, Post Placebo Administration | MUD Group, WT Genotype, Pre Placebo Administration | MUD Group, WT Genotype, Post Placebo Administration | MUD Group, CV Genotype, Pre Methamphetamine Administration | MUD Group, CV Genotype, Post Methamphetamine Administration | MUD Group, WT Genotype, Pre Methamphetamine Administration | MUD Group, WT Genotype, Post Methamphetamine Administration | HC Group, CV Genotype, Pre Placebo Administration | HC Group, CV Genotype, Post Placebo Administration | HC Group, WT Genotype, Pre Placebo Administration | HC Group, WT Genotype, Post Placebo Administration | HC Group, CV Genotype, Pre Methamphetamine Administration | HC Group, CV Genotype, Post Methamphetamine Administration | HC Group, WT Genotype, Pre Methamphetamine Administration | HC Group, WT Genotype, Post Methamphetamine Administration
Number analyzed (Participants) | 7 | 6 | 5 | 5 | 4 | 4 | 7 | 7 | 3 | 3 | 5 | 5 | 4 | 4 | 8 | 8
number of correct answers
  DSST | 42.3 (11.1) | 44.3 (23.3) | 50.8 (3.7) | 53.2 (6.1) | 42.8 (17.2) | 42.5 (9.8) | 42.9 (9.3) | 44.7 (8.8) | 63.7 (8.1) | 57.0 (1.0) | 47.8 (9.1) | 60.4 (15.4) | 75.8 (16.7) | 68.3 (10.0) | 61.0 (9.7) | 59.9 (13.1)
  RVIP | 24.0 (4.4) | 29.7 (8.4) | 29.8 (5.7) | 34.8 (11.5) | 27.5 (13.2) | 33.8 (9.5) | 31.9 (10.0) | 34.3 (7.5) | 28.3 (4.2) | 31.7 (8.1) | 37.8 (9.3) | 39.6 (11.4) | 27.3 (7.8) | 38.3 (5.7) | 35.5 (14.1) | 42.6 (12.3)

5. Secondary Outcome: Methamphetamine Concentration in Saliva (ng/ml)
Description: Saliva samples were acquired to test concentration of methamphetamine levels
Time Frame: 2.5 hours prior to and 3 hours post study drug administration on visits 2 and visit 3 (randomized to placebo or methamphetamine; washout period between visit 2 and 3 was at least 3 days)
Population: Participants were excluded from further analyses if they did not complete all pre and post outcome measures during visit. Placebo and methamphetamine administration include individuals who completed the respective visit at either the first or second intervention. One participant (MUD, CV, post placebo administration) did not complete the final set of data but did complete both imaging measures.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | MUD Group, CV Genotype, Pre Placebo Administration | MUD Group, CV Genotype, Post Placebo Administration | MUD Group, WT Genotype, Pre Placebo Administration | MUD Group, WT Genotype, Post Placebo Administration | MUD Group, CV Genotype, Pre Methamphetamine Administration | MUD Group, CV Genotype, Post Methamphetamine Administration | MUD Group, WT Genotype, Pre Methamphetamine Administration | MUD Group, WT Genotype, Post Methamphetamine Administration | HC Group, CV Genotype, Pre Placebo Administration | HC Group, CV Genotype, Post Placebo Administration | HC Group, WT Genotype, Pre Placebo Administration | HC Group, WT Genotype, Post Placebo Administration | HC Group, CV Genotype, Pre Methamphetamine Administration | HC Group, CV Genotype, Post Methamphetamine Administration | HC Group, WT Genotype, Pre Methamphetamine Administration | HC Group, WT Genotype, Post Methamphetamine Administration
Number analyzed (Participants) | 7 | 6 | 5 | 5 | 4 | 4 | 7 | 7 | 3 | 3 | 5 | 5 | 4 | 4 | 8 | 8
ng/ml | 5320 (4794) | 3750 (3408) | 3328 (3327) | 1827 (1032) | 2828 (1539) | 3140 (3289) | 6067 (8015) | 3984 (3994) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 467 (296) | 0 (0) | 253 (101)

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Methamphetamine: Adverse events related to methamphetamine administration
- Placebo: Adverse events related to placebo administration.
Arm/Group | Methamphetamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 9/24 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methamphetamine (N=24) | Placebo (N=20)
Headache (General disorders) | 2 | 2
Dizziness (General disorders) | 2 | 2
Psychomotor slowing (General disorders) | 0 | 1
Parasthesia (General disorders) | 5 | 1
Confusion/Memory Impairment (General disorders) | 1 | 0
Fatigue/Somnolence (General disorders) | 3 | 1
Taste abnormality (General disorders) | 0 | 1
Dry mouth (General disorders) | 6 | 1
Heart Palpitations (General disorders) | 4 | 0
Other (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03973489/Prot_SAP_000.pdf